CLINICAL TRIAL: NCT03095339
Title: EFECAB: Improving Pig Management to Prevent Epilepsy in Burkina Faso
Acronym: EFECAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: AFRICSanté (Other); Institute of Tropical Medicine, Belgium (Other); Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government); University of Ouagadougou, Burkina Faso (Other); University Hospital, Limoges (Other); Centre Universitaire Souro Sanou (Unknown); Technical University of Munich (Other); Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1419
Record Dates: First submitted 2017-03-22; First posted 2017-03-29 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Cysticercosis
Keywords: Burkina Faso; Community-based randomized controlled trial; Cysticercosis; Implementation Research; Effectiveness
MeSH Terms: conditions — Cysticercosis

STUDY DESIGN:
Intervention Model Description: This is a pre-post community-based randomized controlled trial. The unit of randomization is the village (community)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational package (Active Comparator): The educational package included the offering of the Self-Esteem , Associative strengths, Resourcefulness, Action-planning and Responsibility (SARAR) Participatory Hygiene and Sanitation Transformation (PHAST) approach, a 52 minutes educational movie and accompanying cartoon booklet. The package was developed using the PRECEDE approach.
  Interventions: Other: Educational package
- Control (No Intervention): The control group did not receive any intervention

INTERVENTIONS:
Other: Educational package — The educational package was offered to 30 villages post randomization. The field team completed the SARAR PHAST with community members for 2-3 days in each intervention village. The movie was projected every night for 2-3 days in each intervention village.
  Arms: Educational package

SUMMARY:
This is a pre-post randomized community-based controlled trial aimed at estimating the effectiveness of an educational package developed using PRECEDE PROCEED to reduce the cumulative incidence of Taenia solium cysticercosis in three Provinces of Burkina Faso. The study design included an 18-months baseline study to measure baseline cumulative incidence of cysticercosis followed by an 18-month post randomization study to measure the effectiveness of the intervention. Sixty villages of three Provinces of Burkina Faso were included. The primary outcome was the change in the baseline to post randomization cumulative incidence in the intervention group compared to the control group.

ELIGIBILITY:
The unit of randomization and analysis of this study is the village. Therefore, the eligibility criteria were determined at the village level.

Inclusion Criteria:

* Population of at least 1000 at the 2006 census
* Present on the map of the "Institut Géographique du Burkina 2000"
* Separated from another village by at least 5 kilometers.

Exclusion Criteria:

* Village located on a National or Provincial road
* Village located within 20 km of Koudougou or Ouagadougou
* Regional or Provincial Capital
* Absence of pigs in the village

At the individual level, the following eligibility criteria were used:

Inclusion Criteria:

* Aged 5 years old or more
* Has lived in the village for at least 12 months
* Not planning to move in the next three years

Exclusion Criteria:

* Presence of confirmed epilepsy or progressively worsening severe chronic headaches at baseline.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-02-21 (Actual); Primary Completion 2014-11-24 (Actual); Study Completion 2015-01-31 (Actual)

PRIMARY OUTCOMES:
Human active cysticercosis cumulative incidence | baseline, 18 months follow-up pre randomization, 18 months follow-up post randomization
  Sero conversion to the AgELISA test to detect antigens of cysticercosis

SECONDARY OUTCOMES:
Porcine active cysticercosis prevalence | baseline, 18 months follow-up pre randomization, 18 months follow-up post randomization
  Sero-positivity to the AgELISA test to detect antigens of cysticercosis
Change in knowledge, attitude and practices | baseline, 18 months follow-up pre randomization, 18 months follow-up post randomization
  Change in answers to the questionnaire through time
Cumulative incidence of epilepsy and progressively worsening severe chronic headaches | baseline, 18 months follow-up pre randomization, 18 months follow-up post randomization
  development of neurological disorders among those followed up at least twice
Stigmatization of epilepsy | 18 months follow-up post randomization
  Attitudes and knowledge regarding epilepsy post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Carabin, DVM PhD, Principal Investigator — University of Oklahoma
Locations (1):
- AFRICSanté, Bobo-Dioulasso, Burkina Faso

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available at the time of publication as per NIH requirements

REFERENCES:
- [Background] Carabin H, Traore AA. Taenia solium taeniasis and cysticercosis control and elimination through community-based interventions. Curr Trop Med Rep. 2014 Dec 1;1(4):181-193. doi: 10.1007/s40475-014-0029-4. PMID 25544938
- [Background] Nitiema P, Carabin H, Hounton S, Praet N, Cowan LD, Ganaba R, Kompaore C, Tarnagda Z, Dorny P, Millogo A, Efecab. Prevalence case-control study of epilepsy in three Burkina Faso villages. Acta Neurol Scand. 2012 Oct;126(4):270-8. doi: 10.1111/j.1600-0404.2011.01639.x. Epub 2012 Jan 31. PMID 22289127
- [Background] John CC, Carabin H, Montano SM, Bangirana P, Zunt JR, Peterson PK. Global research priorities for infections that affect the nervous system. Nature. 2015 Nov 19;527(7578):S178-86. doi: 10.1038/nature16033. PMID 26580325
- [Background] Carabin H, Millogo A, Cisse A, Gabriel S, Sahlu I, Dorny P, Bauer C, Tarnagda Z, Cowan LD, Ganaba R. Prevalence of and Factors Associated with Human Cysticercosis in 60 Villages in Three Provinces of Burkina Faso. PLoS Negl Trop Dis. 2015 Nov 20;9(11):e0004248. doi: 10.1371/journal.pntd.0004248. eCollection 2015 Nov. PMID 26588468
- [Background] Dermauw V, Ganaba R, Cisse A, Ouedraogo B, Millogo A, Tarnagda Z, Van Hul A, Gabriel S, Carabin H, Dorny P. Taenia hydatigena in pigs in Burkina Faso: A cross-sectional abattoir study. Vet Parasitol. 2016 Oct 30;230:9-13. doi: 10.1016/j.vetpar.2016.10.022. Epub 2016 Oct 24. PMID 27884445
- [Background] Carabin H, Winkler AS, Dorny P. Taenia solium cysticercosis and taeniosis: Achievements from the past 10 years and the way forward. PLoS Negl Trop Dis. 2017 Apr 20;11(4):e0005478. doi: 10.1371/journal.pntd.0005478. eCollection 2017 Apr. No abstract available. PMID 28426664
- [Result] Ngowi H, Ozbolt I, Millogo A, Dermauw V, Some T, Spicer P, Jervis LL, Ganaba R, Gabriel S, Dorny P, Carabin H. Development of a health education intervention strategy using an implementation research method to control taeniasis and cysticercosis in Burkina Faso. Infect Dis Poverty. 2017 Jun 1;6(1):95. doi: 10.1186/s40249-017-0308-0. PMID 28569208
- [Derived] Sahlu I, Bauer C, Ganaba R, Preux PM, Cowan LD, Dorny P, Millogo A, Carabin H. The impact of imperfect screening tools on measuring the prevalence of epilepsy and headaches in Burkina Faso. PLoS Negl Trop Dis. 2019 Jan 17;13(1):e0007109. doi: 10.1371/journal.pntd.0007109. eCollection 2019 Jan. PMID 30653519
- See also: Website of the facility in Burkina Faso which managed the study — http://africsante.org/

DOCUMENTS (1):
  • Study Protocol (2014-10-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT03095339/Prot_000.pdf